CLINICAL TRIAL: NCT01693159
Title: Randomized Controlled Multicenter Trial to Evaluate the Effects of Ethyl-2-cyanoacrylate on Pain Intensity and Quality of Life in Head and Neck Cancer Patients Suffering From Cetuximab-induced Rhagades During Radioimmunotherapy
Brief Title: Effects of ECA on Quality of Life in Head and Neck Cancer Patients Suffering From Cetuximab-induced Rhagades
Acronym: SUPPORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: Heidelberg University (Other); iOMEDICO AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Uni-HD-2010-33-40-1003
Record Dates: First submitted 2012-09-18; First posted 2012-09-26 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Pain
Keywords: Painful cetuximab-induced rhagades; Radioimmunotherapy; Head and neck cancer
MeSH Terms: conditions — Pain; Head and Neck Neoplasms | interventions — Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECA: Ethyl-2-cyanoacrate (Experimental): Application of ethyl-2-cyanoacrylate (ECA) for painful cetuximab-induced rhagades
  Interventions: Device: ECA
- Standard treatment of the institution (Active Comparator): Standard treatment of the institution to treat painful cetuximab-induced rhagades
  Interventions: Other: Standard topical treatment of the institution, e.g. Lotio

INTERVENTIONS:
Device: ECA — In the experimental arm patients will be topically treated with the liquid glue ethyl-2-cyanoacrylate (ECA).
  Other Names: Ethyl-2-cyanoacrylate (ECA)
  Arms: ECA: Ethyl-2-cyanoacrate
Other: Standard topical treatment of the institution, e.g. Lotio — Standard treatment of the institution to treat painful cetuximab-induced rhagades
  Other Names: Ointment, Creme, Lotio, for example dexpanthenol-containing topical treatment
  Arms: Standard treatment of the institution

SUMMARY:
The SUPPORT trial is an open-label, prospective, randomized, national multicenter intervention study to evaluate the effectiveness of ethyl-2-cyanoacrylate versus the standard treatment of each institution on the pain intensity and QoL in patients with locally advanced head and neck cancer suffering from painful cetuximab-induced rhagades during radioimmunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced squamous cell carcinoma of the head and neck and participation in the HICARE-phase-IV-trial
* Cetuximab-induced painful rhagades, i.e. SUPO Score 2-3 (see Figure 2)
* Compliance to the photo documentation
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Cetuximab-induced rhagades without any pain, i.e. SUPO Score 1
* Cetuximab-induced rhagades, SUPO Score 4, i.e. superinfection of the rhagades
* Patients not being enrolled in the HICARE trial
* Substance misuse, psychoactive substance abuse or psychological/social conditions leading to a decreased patients' compliance with possible bad influence to the results of the study
* Known allergic reaction to ethyl-2-cyanoacrylate (ECA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2018-07 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
pain intensity 24 hours after application of ECA or the standard treatment quantified by the visual analogue scale (VAS) | 24 hours after application
  pain intensity quantified by the visual analogue scale (VAS)

SECONDARY OUTCOMES:
Evaluation of QoL | 5 to 7 days after application of treatment
  Evaluation of QoL assessed by the EORTC-QoL-C30 questionnaire and the Dermatological Life Quality Index (DLQI)

OTHER OUTCOMES:
SUPO-Score for classification of cetuximab-induced rhagades | 24 hours and 5 to 7 days after application of treatment
  SUPO-Score for classification of cetuximab-induced rhagades:
  Grade 1: Rhagades without clinical symptoms
  Grade 2: Painful rhagades Grade 2a: Moderate pain, no impairment of activity in the daily routine (ADL) Grade 2b: Severe pain and impairment of the activities of daily living (ADL) Grade 3: Painful, deep and spontaneously bleeding rhagades
  Grade 4: Superinfection of the rhagades (detection of bacterial growth) Grade 4a: Local infection Grade 4b: Systemic infection
  Grade 5: Death due to complications of the rhagades
Adverse Events of ECA | from time of randomization untio end of study, i.e. until 5 to 7 days after application of treatment
  Adverse Events of ECA due to NCI CTCAE v. 4.02

CONTACTS AND LOCATIONS:
Overall Officials: Karin Potthoff, MD, Principal Investigator — National Center for Tumor Diseases, Heidelberg
Locations (1):
- University of Heidelberg Medical Center, Heidelberg, Germany

REFERENCES:
- [Derived] Potthoff K, Habl G, Bruckner T, Suppan C, Hassel J, Jager D, Indorf M, Debus J. Randomized controlled trial to evaluate the effects of ethyl-2-cyanoacrylate on pain intensity and quality of life in head and neck cancer patients suffering from cetuximab-induced rhagades during radioimmunotherapy: the support trial. BMC Cancer. 2014 Apr 17;14:270. doi: 10.1186/1471-2407-14-270. PMID 24742019